CLINICAL TRIAL: NCT02497924
Title: A Phase 1 Study to Investigate Absorption, Metabolism, and Excretion After Establishment of Steady State Via GBT440 Loading and Maintenance Dosing Followed by a Single Oral Dose Administration of [14C]-GBT440 in Healthy Male Subjects
Brief Title: A Study of the Absorption, Metabolism, and Excretion of GBT440 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Blood Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GBT440-002
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2015-09

CONDITIONS: Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GBT440 (Experimental): GBT440 / [C14] GBT440
  Interventions: Drug: GBT440

INTERVENTIONS:
Drug: GBT440 — GBT440 capsules followed by single dose of [C14] GBT440 oral suspension

SUMMARY:
This study will provide information regarding the metabolic pathway of GBT440, the need for evaluation of potential drug-drug interactions, and the need for studies in special populations. The administration of radiolabeled drug is necessary to fully characterize the rates and routes of elimination of GBT440, providing further quantitative information on the disposition of GBT440. The results from this study will permit a comprehensive comparison between animal and human routes of elimination and metabolic profiles of GBT440.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy; non-smoking male; 18 to 55 years old, inclusive
2. Weighs at least 50 kg and not more than 110 kg
3. Agrees to use contraception
4. Willing and able to give written informed consent

Exclusion Criteria:

1. Evidence or history of clinically significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
2. History of stomach or intestinal surgery that would potentially alter drug absorption
3. History of hypersensitivity or allergy to drugs, foods, or other substances
4. History or presence of abnormal electrocardiogram
5. Exposure to significant radiation or participated in more than 1 other radiolabeled study drug trial within 12 months of Screening
6. Participated in another clinical trial of an investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to Screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Area under the whole blood and plasma concentration versus time curve (AUC) | 0 to 648 hours post dose
Peak whole blood and plasma concentration (Cmax) | 0 to 168 hours post dose
Time to peak whole blood and plasma concentration (Tmax) | 0 to 168 hours post dose
Half-life (T 1/2) | 0 to 168 hours post dose
Percent total recovery of radioactivity in blood, urine, and feces | 0 to 648 hours post dose
Identification of metabolites in whole blood, plasma, urine, and feces following [C14] GBT440 administration | 0 to 168 hours post dose

SECONDARY OUTCOMES:
Number of participants with adverse events | Baseline to 27 days

CONTACTS AND LOCATIONS:
Overall Officials: Carla Washington, PhD, Study Director — Global Blood Therapeutics
Locations (1):
- Covance Early Clinical Services, Madison, Wisconsin, United States